CLINICAL TRIAL: NCT06530706
Title: Effect of Esketamine on Anxiety State in Patients Undergoing Abdominal Tumor Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, attending, principle investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-2024-327（IIT）
Record Dates: First submitted 2024-07-29; First posted 2024-07-31 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Anxiety State; Esketamine
Keywords: esketamine; anxiety state
MeSH Terms: conditions — Anxiety Disorders | interventions — Esketamine; Saline Solution; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiment group (Experimental): Esketamine 0.2mg/kg was given slowly after intubation, and then 0.1mg/kg/h was pumped continuously until the end of the operation. Patients received sufentanil based patient-controlled intravenous analgesia (PCIA) within 72 hours postoperatively, with sufentanil combined with esketamine 1mg/kg in a PCIA device.
  Interventions: Drug: Esketamine
- Control group (Placebo Comparator): Same volume of normal saline was given slowly after intubation, and then pumped continuously until the end of the operation. Patients received sufentanil based patient-controlled intravenous analgesia (PCIA) within 72 hours postoperatively, without esketamine in the PCIA device.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Esketamine — Esketamine 0.2mg/kg was pumped slowly after intubation, followed by 0.1mg/kg pumped until the end of the operation. In the PCIA pump, esketamine 1mg/kg was added to the sufentanil.
  Other Names: Experimental group
  Arms: Experiment group
Drug: normal saline — Same volume of normal saline was pumped slowly after intubation, followed by the same volume of NS until the end of the operation. In the PCIA pump, only sufentanil was used.
  Other Names: Control Group
  Arms: Control group

SUMMARY:
To evaluate whether esketamine can relieve anxiety in patients undergoing abdominal tumor surgery.

DETAILED DESCRIPTION:
Hamilton anxiety Scale was used to screen patients with anxiety. Only patients with score ≥ 8 were enrolled. These patients were randomly assigned to the experimental group and control group.

All patients enrolled were evaluated with Hamilton anxiety Scale, PHQ-8 scale, QoR-15 Scale and Athens Insomnia Scale. After induction, sevoflurane and remifentanil were used to maintain anesthesia. The experimental group had esketamine while the control group had normal saline. Athens Insomnia Scale was used to assess the sleep status 1, 2, 3 days after surgery and 1 month after surgery. Hamilton anxiety Scale was used to evaluate the anxiety state of the patients 3 days after surgery and 1 month after surgery. PHQ-8 scale, QoR-15 Scale were collected 3 days after surgery and 1 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominal tumor surgery;
* older than 18 years old and younger than 70 years old;
* ASA grade I-III；
* Hamilton anxiety scale ≥ 8.

Exclusion Criteria:

* Having serious mental illness before surgery or on antipsychotic medication in the two weeks before screening;
* Severe organ function lesions such as heart failure (left ventricular ejection fraction <30%), myocardial infarction, kidney failure (requiring kidney replacement therapy), liver function impairment (Child-Pugh grade C), etc.
* Patients arranged to receive general anesthesia combined with epidural anesthesia patients;
* Patients who cannot communicate, read or write due to visual, auditory, language or other reasons;
* Patients allergic to ketamine;
* Patients refused to use postoperative self-controlled intravenous analgesia pump;
* Patients refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Whether esketamine can reduce anxiety status in patients with anxiety | 1 day before surgery, 3 days after surgery, 1 month after surgery
  assessed by Hamilton anxiety scale. The score ranges from 0 to 56, while the higher score means a more anxious state.

SECONDARY OUTCOMES:
To explore whether esketamine can improve sleep status | 1 day before surgery, 1,2 and 3 days after surgery, 1 month after surgery
  assessed by Athens Insomnia Scale. Athens Insomnia Scale ranges from o to 24, with a higher score means a worse sleep status.
To explore whether esketamine can improve life quality | 1 day before surgery, 3 days after surgery, 1 month after surgery
  assessed by QoR-15 (quality of recovery-15). The score ranges from 0 (bad quality) to 150 (good quality).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang cancer hospital, Hangzhou, Zhejiang, China